CLINICAL TRIAL: NCT07045688
Title: Efficacy of Vonoprazan Based Dual and Triple Therapy for Naive Patient With Helicobacter Pylori Infection
Brief Title: Efficacy of Vonoprazan Based Dual and Triple Therapy for Patient With Helicobacter Pylori Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Andrew Kamil Wadie, Resident,Internal Medicine Departement , Faculty of Medicine Sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-5-10MS
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Efficacy of Vonoprazan based dual therapy for naive patient with Helicobacter Pylori infection (Active Comparator): we assess the efficacy of Vonoprazan based dual therapy for eradication of Helicobacter Pylori infection in naive patient.
  Interventions: Drug: Efficacy of Vonoprazan based dual therapy for naive patient with Helicobacter Pylori infection
- Efficacy of Vonoprazan based triple therapy for naive patient with Helicobacter Pylori infection (Active Comparator): we assess the efficacy of Vonoprazan based triple therapy for eradication of Helicobacter Pylori infection in naive patient.
  Interventions: Drug: Efficacy of Vonoprazan based triple therapy for naive patient with Helicobacter Pylori infection
- Efficacy of PPI based triple therapy for naive patient with Helicobacter Pylori infection (Active Comparator): we assess the efficacy of proton pump inhibitors (PPI) based dual therapy for eradication of Helicobacter Pylori infection in naive patient.
  Interventions: Drug: Efficacy of PPI based triple therapy for naive patient with Helicobacter Pylori infection

INTERVENTIONS:
Drug: Efficacy of Vonoprazan based dual therapy for naive patient with Helicobacter Pylori infection — we assess the efficacy of Vonoprazan based dual therapy for eradication of Helicobacter Pylori infection in naive patient.
  Arms: Efficacy of Vonoprazan based dual therapy for naive patient with Helicobacter Pylori infection
Drug: Efficacy of Vonoprazan based triple therapy for naive patient with Helicobacter Pylori infection — we assess the efficacy of Vonoprazan based triple therapy for eradication of Helicobacter Pylori infection in naive patient.
  Arms: Efficacy of Vonoprazan based triple therapy for naive patient with Helicobacter Pylori infection
Drug: Efficacy of PPI based triple therapy for naive patient with Helicobacter Pylori infection — we assess the efficacy of PPI based triple therapy for eradication of Helicobacter Pylori infection in naive patient.
  Arms: Efficacy of PPI based triple therapy for naive patient with Helicobacter Pylori infection

SUMMARY:
This study aims to assess Efficacy of vonoprazan based dual and triple therapy for naïve patient with Helicopacter Pylori infection in Sohag Government .

ELIGIBILITY:
Inclusion Criteria:

* Age: >18 years old.
* H. pylori infection: Confirmed by histopathology or non-invasive tests (e.g., stool antigen test).

Exclusion Criteria:

* Prior H. pylori treatment: Previous treatment for H. pylori infection.
* Allergies: Known allergies to study medications or components.
* Patients cannot finish treatment course.
* Patient missed follow up.
* Patients refusing or neglecting test of cure for H. pylori.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
efficacy medical treatment for eradication of Helicobacter Pylori infection in naive patient. | 4 weeks after successful medical treatment
  stool antigen for H. Pylori

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Background] Chey WD, Leontiadis GI, Howden CW, Moss SF. ACG Clinical Guideline: Treatment of Helicobacter pylori Infection. Am J Gastroenterol. 2017 Feb;112(2):212-239. doi: 10.1038/ajg.2016.563. Epub 2017 Jan 10. PMID 28071659
- [Background] Argueta EA, Alsamman MA, Moss SF, D'Agata EMC. Impact of Antimicrobial Resistance Rates on Eradication of Helicobacter pylori in a US Population. Gastroenterology. 2021 May;160(6):2181-2183.e1. doi: 10.1053/j.gastro.2021.02.014. Epub 2021 Feb 9. No abstract available. PMID 33577874